CLINICAL TRIAL: NCT07260500
Title: A Phase II, Multicenter, Randomized, Open-label, Active-controlled Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of Polyethylene Glycol Recombinant Human Growth Hormone Injection in Short Children Born Small for Gestational Age (SGA)
Brief Title: A Phase II Study of PEG-rhGH Injection for Short Children Born Small for Gestational Age: Efficacy, Safety, and Pharmacokinetics
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GenSci031-202
Record Dates: First submitted 2025-11-21; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Short Stature Children Born Small for Gestational Age (SGA)
MeSH Terms: interventions — polyethylene glycol-recombinant human growth hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PEG-rhGH dose 1 weekly (Experimental): Jintrolong® dose 1, subcutaneous injection, once every week for 26 weeks.
  Interventions: Drug: PEG-rhGH Injection
- PEG-rhGH dose 2 weekly (Experimental): Jintrolong® dose 2, subcutaneous injection, once every week for 26 weeks
  Interventions: Drug: PEG-rhGH Injection
- Daily hGH (active control) (Active Comparator): Jintropin® dose 3, subcutaneous injection, once daily for 26 weeks.
  Interventions: Drug: hGH Injection

INTERVENTIONS:
Drug: PEG-rhGH Injection — Jintrolong® Dose 1, subcutaneous injection, once weekly for 26 weeks for 24 subjects..
  Jintrolong® Dose 2, subcutaneous injection, once weekly for 26 weeks for 24 subjects..
  Other Names: Jintrolong®
  Arms: PEG-rhGH dose 1 weekly; PEG-rhGH dose 2 weekly
Drug: hGH Injection — Jintropin® dose 3, subcutaneous injection, once daily for 26 weeks (active comparator) for 24 subjects.
  Other Names: Jintropin®
  Arms: Daily hGH (active control)

SUMMARY:
This study will take place at multiple sites and is divided into three phases:an initial 4-week getting-to-know-you phase,a 26-week main phase where participants receive medication,and a 4-week follow-up phase.Participants will be divided into three groups:two will receive different doses of PEG-rhGH Injection,and the third will receive hGH Injection.The goal is to determine which medication works best.

ELIGIBILITY:
Inclusion Criteria:

* Born full-term and "small-for-dates" - Born at 37-41 weeks (full-term). - Birth weight below the 10th percentile for that week of pregnancy and sex .
* At least 3 years old on the day the parent signs the consent form.
* Still prepubertal (Tanner stage I - no signs of puberty yet).
* Height at the first study visit is more than 2 standard deviations below the average for his or her age and sex.
* Bone age on X-ray is no more than 1 year ahead of real age.
* Never taken growth hormone, IGF-1, or any ghrelin-like medicine before.
* Child and parent/guardian are willing to sign the consent form and follow the study visits.

Exclusion Criteria:

* Severe allergy to growth hormone or its ingredients.
* Growth-hormone deficiency.
* Any chromosome/genetic/syndrome cause of short stature.
* Other diseases that can impair growth.
* Cognitive, developmental, or psychiatric disorders that could affect assessments .
* Current or past cancer, or high familial cancer risk.
* Positive hepatitis B, hepatitis C, HIV, or active tuberculosis at screening.
* Abnormal liver or kidney blood tests.
* Pre-diabetes or diabetes at screening .
* Systemic steroids > 28 consecutive days or > 14 days total in the last 3 months.
* High-dose inhaled steroids > 28 days in the last year.
* Prior use of aromatase inhibitors, GnRH analogues, sex hormones, anabolic agents, or other drugs that affect growth. 13. Unable to receive subcutaneous injections.
* Claustrophobia or inability to undergo brain MRI.
* Participated in another clinical trial with investigational treatment within 3 months.
* Any other condition that, in the investigator's opinion, makes the child unsuitable for the study.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-11-11 (Actual); Primary Completion 2026-10-26 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Annual height velocity at Week 26 of treatment | 26 Weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital Affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei, China